CLINICAL TRIAL: NCT05950061
Title: Sertraline Versus Escitalopram in South Asian Participants With Moderate to Severe Major Depressive Disorder: A Double-blind, Parallel, Randomized Controlled Trial
Brief Title: Sertraline Versus Escitalopram in South Asian Participants With Moderate to Severe Major Depressive Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: KRL Hospital, Islamabad (Other)
Collaborators: Khyber Medical College, Peshawar (Other); Quaid-e-Azam Medical College (Other); Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Hassan Mumtaz, Principal Researcher, KRL Hospital, Islamabad
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KRL/02/19/1
Record Dates: First submitted 2023-06-30; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder
Keywords: Sertraline; Depressive Disorder, Major; Escitalopram; South Asian People; Humans
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Sertraline; Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sertraline (Experimental): Sertraline
  Interventions: Drug: Sertraline
- Escitalopram (Experimental): Escitalopram
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Sertraline — Sertraline (200 mg/day) capsule
  Other Names: Sertraline pill
  Arms: Sertraline
Drug: Escitalopram — Escitalopram (10 mg/day) capsule
  Other Names: Escitalopram pill
  Arms: Escitalopram

SUMMARY:
Objective: The aim of this randomized controlled trial was to compare the efficacy and safety of sertraline and escitalopram in participants with moderate to severe major depressive disorder (MDD).

Methods: A total of 744 participants with moderate to severe MDD were randomly assigned to receive either sertraline or escitalopram for 8 weeks. Drug dosages and titration schedules were based on the recommendations of the prescribing information for each product and according to the judgment of the clinicians involved in the study.

The primary outcome measures were changes from baseline on the Montgomery-Åsberg Depression Rating Scale (MADRS) and the Clinical Global Impression (CGI) scale as well as frequency of adverse events in both groups.

DETAILED DESCRIPTION:
This is a monocentric, double-blind, parallel, randomized controlled trial conducted in Khan Research Laboratories (KRL) hospital, Islamabad, Pakistan for a total period of 16 weeks. By employing appropriate measures to ensure adequate allocation concealment, thereby minimizing the potential for selection bias in the assignment of participants to treatment groups, the investigators studied if there was any significant difference in in efficacy and tolerability of oral sertraline (50 - 200 mg/day) and oral escitalopram (10 mg/day) given either at night or during the day in the South Asian population for the treatment of moderate to severe major depressive disorder (MDD). 744 South Asian patients with moderate to severe MDD as per the Montgomery-Asberg Depression Rating Scale (MADRS) scale who had consented to participate in the trial and who fulfilled the inclusion criteria were included in our study. The study was conducted at KRL hospital.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants had to have a score of at least 20 on the MADRS at both screening and baseline visits.
* All participants who had moderate or severe depression
* Study participants had to have normal results on physical examination, laboratory tests, and electrocardiograms, or any abnormalities had to be clinically insignificant.
* Female participants of childbearing potential had to have a negative pregnancy test and be using medically approved contraception.

Exclusion Criteria:

* Lactating women were not eligible to participate.
* Individuals with a psychiatric disorder other than MDD
* Individuals with a history of any Diagnostic and Statistical Manual -V defined psychotic disorder
* Individuals with current diagnosis of bipolar disorder
* Individuals with current diagnosis of schizophrenia
* Individuals with current diagnosis of obsessive-compulsive disorder
* Individuals with intellectual disability
* Individuals with a pervasive development disorder.
* Participants with current substance abuse or dependency,
* Participants with suicidal risk,
* Participants with personality disorders that would impede participation in study
* Participants were also not eligible to participate if they had used a selective serotonin release inhibitor (SSRI) in the past two weeks (past five weeks if they used fluoxetine).
* Participants with Montgomery-Åsberg Depression Rating Scale score of <19.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2023-02-26 (Actual)

PRIMARY OUTCOMES:
Change in clinical global impression (CGI) scale | 4 months
  Change in the clinical global impression scale. CGI is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill)
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) scale | 4 months
  Change in Montgomery-Åsberg Depression Rating Scale from baseline. The MADRS (Montgomery & Åsberg, 1979) comprises the following 10 items: apparent sadness; reported sadness; inner tension; reduced sleep; reduced appetite; concentration difficulties; lassitude; inability to feel; pessimistic thoughts; and suicidal thoughts. Clinicians rate each item on a 7-point Likert scale; the sum of the item scores produces a MADRS total score that ranges from 0 to 60, with higher scores reflecting greater depression severity.
Diarrhea | 4 months
  Number of participants with diarrhea
Nausea | 4 months
  Number of participants with nausea
Sexual dysfunction | 4 months
  Number of participants with sexual dysfunction
Upper respiratory tract infection | 4 months
  Number of participants with upper respiratory tract infection

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Mumtaz, MBBS, MRSPH, Study Director — KRL Hospital, Islamabad
Locations (1):
- KRL Hospital, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided